CLINICAL TRIAL: NCT03836274
Title: Tolerance and Acceptability Evaluation of MONACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aymes International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AY:ASK-SCH
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients established on an oral nutritional supplement (ONS), requiring nutritional supplementation of at least 300kcal/day will be changed onto an equivalent prescription of AYMES 'MONACO' for a period of 9 days.
  Interventions: Dietary Supplement: AYMES MONACO

INTERVENTIONS:
Dietary Supplement: AYMES MONACO — AYMES MONACO is a Food for Special Medical Purposes (FSMP) and must, therefore, be used under medical supervision. It is not designed as a sole source of nutrition.

SUMMARY:
To evaluate tolerance and acceptability of 'MONACO' in patients requiring supplementary oral nutritional support compared with currently available alternatives.

DETAILED DESCRIPTION:
To evaluate tolerance and acceptability of 'MONACO' in patients requiring supplementary oral nutritional support compared with currently available alternatives, measuring outcomes of GI effects, Compliance, product preference, convenience etc.

To obtain data to support an ACBS submissions for 'MONACO' (to allow for prescription in the community at NHS expense).

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years) who are able to communicate clearly.
* Patients with or at risk of malnutrition as determined by growth charts and/or by professional clinical judgement.
* Patients expected to require oral nutritional supplementation for at least 2 further weeks.
* Patients requiring supplementary intake approximately 300 kcal /day from an oral nutritional supplement
* Informed assent/consent obtained.

Exclusion Criteria:

* Patients with cow's milk protein allergy requiring a milk free diet
* Patients with inherited metabolic conditions.
* Patients requiring enteral tube feeding or parenteral nutrition.
* Patients with medical or dietary contraindication to any feed ingredients (see appendix 2 for full ingredient list)
* Patients with significant renal (requiring dialysis) or hepatic impairment (e.g. hepatitis)
* Patients with dysphagia requiring stage 1, 2 or 3 thickened fluids.
* Patients with uncontrolled inflammatory bowel disease or previous bowel resection with ongoing gastrointestinal symptoms.
* Patients for whom the investigator has concerns regarding the ability or willingness of the patient and or carer to comply with protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within 2 weeks prior to entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
GI Tolerance | 9 Days
  To assess gastro-intestinal tolerance of 'MONACO' in patients in the community requiring oral nutritional supplementation. Monitoring includes recording the number and consistency of bowel movements, any episodes of nausea, vomiting, abdominal pain, bloating or diarrhoea.

SECONDARY OUTCOMES:
Acceptability and Palatability of Consuming the Nutritional Supplement: questionnaire | 9 days
  To assess the acceptability of 'MONACO' in patients in the community requiring oral nutritional supplementation. At the end of the intervention period an acceptability and preference questionnaire will be completed by the patient in order to seek their opinion on the taste, smell, texture and overall liking of the new supplement drink. A 5 point hedonic scale will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- AYMES International, Haywards Heath, United Kingdom

IPD SHARING:
Plan to Share IPD: No